CLINICAL TRIAL: NCT01775462
Title: A Phase 2 Open-label, Dose-escalation Study to Evaluate the Safety, Pharmacokinetics, Immunogenicity and Pharmacodynamics/Efficacy of EDI200, an EDA-A1 Replacement Protein, Administered to Male Infants With X-Linked Hypohidrotic Ectodermal Dysplasia (XLHED)
Brief Title: Phase 2 Study to Evaluate Safety, Pharmacokinetics, Immunogenicity and Pharmacodynamics/Efficacy of EDI200 in Male Infants With X-Linked Hypohidrotic Ectodermal Dysplasia (XLHED)
Acronym: ECP-002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Edimer Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECP-002
Record Dates: First submitted 2013-01-17; First posted 2013-01-25 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: X-Linked Hypohidrotic Ectodermal Dysplasia
Keywords: Hypohidrotic Ectodermal Dysplasia; XLHED
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic | interventions — Fc-EDA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EDI200, 3mg/kg (Experimental): Five doses of EDI200 given at 3 mg/kg twice weekly
  Interventions: Drug: EDI200
- EDI200, 10 mg/kg (Experimental): Five doses of EDI200 given at 10 mg/kg twice weekly
  Interventions: Drug: EDI200

INTERVENTIONS:
Drug: EDI200 — 3 or 10 mg/kg of EDI200
  Other Names: APO200

SUMMARY:
This Phase 2 first-in-neonate EDI200 study will enroll treatment-naïve, XLHED-affected male newborns in the first two weeks of life. All subjects will meet entry criteria including documentation of an Ectodysplasin (EDA) mutation associated with XLHED. Following Baseline evaluations, EDI200 dosing will be initiated between day-of-life 2 and 14, with each study subject receiving 2 doses/week for a total of 5 doses. The study will enroll subjects in two cohorts with subjects in cohort 1 dosed at 3 mg/kg/dose, associated with partial efficacy, and cohort 2 dosed at 10 mg/kg/dose where enhanced efficacy was demonstrated in the most relevant preclinical model. Given the challenge of identifying families where the subject is yet to be born, it is expected that cohort size and time for recruitment will be variable.

DETAILED DESCRIPTION:
This Phase 2 first-in-neonate EDI200 study will enroll treatment-naïve, XLHED-affected male newborns in the first two weeks of life. All subjects will meet entry criteria including documentation of an EDA mutation associated with XLHED. Following Baseline evaluations, EDI200 dosing will be initiated between day-of-life 2 and 14, with each study subject receiving 2 doses/week for a total of 5 doses. This dosing regimen mirrors that used to enhance efficacy in the dog XLHED model, considered to be most relevant to the clinical study design. The study will enroll subjects in two cohorts with subjects in cohort 1 dosed at 3 mg/kg/dose, associated with partial efficacy, and cohort 2 dosed at 10 mg/kg/dose where enhanced efficacy was demonstrated in the most relevant preclinical model. Given the challenge of identifying families where the subject is yet to be born, it is expected that cohort size and time for recruitment will be variable. The sponsor anticipates enrollment and dosing of 6-10 subjects over a 12-18 month period, 3-5 subjects per cohort.

ELIGIBILITY:
Inclusion Criteria:

Subjects for study drug administration must meet all of the following criteria to be enrolled:

1. Male with genetic confirmation of an XLHED diagnosis.
2. Subject must be at least 48 hours age and no older than 14 days.
3. Subject will have reached term (defined as 37 weeks gestation or older) prior to receiving first dose study drug.
4. Written informed consent of both parents (if reasonably available) must be obtained for treatment of their XLHED-affected male infant.
5. Neither mother nor the XLHED-affected male infant known to have received an investigational study drug in the 9 months prior to study subject enrollment in this study.
6. No major medical issues that the PI considers a contraindication to participation.

Siblings of subjects receiving study drug must meet all of the following criteria to be enrolled in the natural history sub-study (no age limit involved):

1. Provide written informed consent/assent.
2. A full or half-sibling of a study subject where the study subject has received at least one dose of study drug in the Phase 2 XLHED Neonate Study and has not yet completed the study.
3. No major medical issues that the investigator considers contraindications to participation.

Exclusion Criteria:

Subjects for study drug administration who meet any of the following criteria cannot be enrolled in this study:

1. Medically significant postnatal complications or congenital anomalies outside of those considered to be associated with the diagnosis of XLHED.

Siblings of subjects receiving study drug who meet any of the following criteria cannot be enrolled in the natural history sub-study:

1. Known hypersensitivity to pilocarpine or pilocarpine-like muscarinic agonists.
2. Known hypersensitivity to lidocaine or lidocaine-like agents.
3. Presence of pacemaker.
4. Subjects who are not able or are not willing to comply with the procedures of this protocol.
5. Subject has a condition, which in the opinion of the investigator would not allow for safe conduct of the study.

Ages: 48 Hours to 14 Days | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Up to 6 months after dosing
To assess the antibody response to EDI200 | Up to 6 months after dosing
Area under the concentration time curve to the end of the dosing period (AUC0-tau) of EDI200 | Pre-dose and 15 minutes and 3, 8, 24 and 48 hours post-dose 1 and pre-dose and 15 minutes and 3, 18, 48 and 168 hours post-dose 5
Peak plasma concentration (Cmax) of EDI200 | Pre-dose and 15 minutes and 3, 8, 24 and 48 hours post-dose 1 and pre-dose and 15 minutes and 3, 18, 48 and 168 hours post-dose 5
Time at which maximum concentration is observed (Tmax) of EDI200 | Pre-dose and 15 minutes and 3, 8, 24 and 48 hours post-dose 1 and pre-dose and 15 minutes and 3, 18, 48 and 168 hours post-dose 5

SECONDARY OUTCOMES:
To assess the pharmacodynamics/efficacy (growth and development) of EDI200 | Baseline and 2, 4 and 6 months
To assess the pharmacodynamics/efficacy (dentition) of EDI200 | Baseline and post-six months (extension study)
To assess the pharmacodynamics/efficacy (craniofacial development) of EDI200 | Baseline and 6 months
To assess the pharmacodynamics/efficacy (sweat duct density) of EDI200 | Baseline and 2 and 6 months
To assess the pharmacodynamics/efficacy (sweat rate) of EDI200 | Baseline and 2 and 6 months
To assess the pharmacodynamics/efficacy (Dry eye signs and symptoms) of EDI200 | Baseline and 2 and 6 months
To assess the pharmacodynamics/efficacy (thermoregulation) of EDI200 | Baseline and study day 21
To assess the pharmacodynamics/efficacy (molecular expression profile of skin biopsy tissue) of EDI200 | Baseline, study days 1 and 15

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Huttner, MD, PhD, Study Director — Edimer Pharmaceuticals
Locations (7):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Washington University School of Medicine, St Louis, Missouri
- Hôpital Necker-Enfants Malades, Paris, France
- University Hospital Erlangen, Erlangen, Bavaria, Germany
- Azienda Ospedaliera-Polo Universitario "Luigi Sacco", Milan, Italy
- University Hospital of Wales, Cardiff, United Kingdom

REFERENCES:
- See also: Sponsor's website — http://www.edimerpharma.com